CLINICAL TRIAL: NCT03239509
Title: 15 Years Outcomes Following Bioprosthetic vs Mechanical Isolated Aortic Valve Replacement for Aortic Stenosis in Patients Aged 50 to 65 Years in South Spain. The Andalousian Aortic Valve Multicentric Study (ANDALVALVE)
Brief Title: 15 Years Outcomes Following Bioprosthetic vs Mechanical Aortic Valve Replacement Between 50-65 Years
Acronym: ANDALVALVE
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Other Study IDs: ANDALVALVE STUDY
Record Dates: First submitted 2017-07-12; First posted 2017-08-04 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-01

CONDITIONS: Surgery; Survival, Prosthesis; Valve Heart Disease
Keywords: long-term survival; bioprosthesis; complications; anticoagulation; mechanichal prosthesis
MeSH Terms: conditions — Prosthesis Failure; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bioprosthesis: All patients operated on of isolated AVR with a bioprosthesis implantation between 2000-2015 and age 50-65 years both inclusive.
  Interventions: Procedure: bioprosthesis implantation between 2000-2015
- Mechanical prosthesis: All patients operated on of isolated AVR with a Mechanical prosthesis implantation between 2000-2015 and age 50-65 years both inclusive.
  Interventions: Procedure: mechanical prosthesis implantation between 2000-2015

INTERVENTIONS:
Procedure: bioprosthesis implantation between 2000-2015 — Implantation of a bioprosthesis in aortic position with cardiopulmonary bypass
  Groups: Bioprosthesis
Procedure: mechanical prosthesis implantation between 2000-2015 — Implantation of a mechanical prosthesis in aortic position with cardiopulmonary bypass
  Groups: Mechanical prosthesis

SUMMARY:
Currently there is an increase in the use of bioprosthesis worldwide (> 70% according to national data of the Spanish Society of Thoracic and Cardiovascular Surgery).

There is conflicting evidence regarding the long-term survival of patients aged 50-65 years with mechanical (M) or biological (B) aortic prostheses. General consensus of greater complications associated with the use of long-life anticoagulation in M and of reoperation in B.

Similar survival with lower MACCE complications in bioprosthesis could reconsider their choice in patients aged 50-65 years, specially in the current TAVI era.

The investigators are going to perform a multicentric retrospective observational study (Registry) about 15 year-outcomes Following Bioprosthetic vs Mechanical Isolated Aortic Valve Replacement for Aortic Stenosis in Patients Aged 50 to 65 Years in 5 Cardiovascular Surgery Centers in Andalousia (south Spain)

DETAILED DESCRIPTION:
Objectives The main objective is to analyze long-term survival (15 years) and major cardiovascular complications (MACE, (death of any cause, neurological events (TIA / stroke), any prosthesis reoperation, and major bleeding), in patients aged 50-65 years who underwent isolated aortic valve replacement (AVR) due to severe aortic stenosis . Secondary objectives were to analyze the evolution of transprosthetic gradients by echocardiography, type of INR control, and degree of significant structural degeneration in bioprostheses.

Material and Method: A retrospective analytical study of patients aged 50-65 years who underwent AVR surgery for stenosis between 2000-2015 in all centers with a Cardiovascular Surgery Dept. in Andalousia (SPAIN) as an inclusion criterion. As exclusion criteria, autonomic change of residence, need for concomitant surgery, previous cardiac interventions and endocarditis. Survival analysis and clinical data will be performed through the Diraya Health Care medical records (DAE), direct telephone contact with family and / or relatives, A crude analysis of the data and a posterior analysis by propensity score matching with the help of the Foundation for Biomedical Research of Malaga (IBIMA) with SPSS software will be carried out using a 1: 1 "nearest neighbour" matching protocol based on the Number of total bioprosthesis. A total sample of more than 1200 cases is expected, of which about 380 would be bioprostheses that would serve as a basis for the pairing. To find a 10% difference in the primary endpoint, two groups of 325 patients are required for a p = 0.05 and 80% for a bilateral contrast of two independent proportions. Sub-analysis will be performed by subgroups of age (50-59 vs. 60-65 years) and another according to the mark of the 2 prostheses of each type most used. All statistical analyzes will be two-tailed with an alpha error of 0.05 to consider statistically significant data, and will be reviewed by IBIMA biostatistics.

Conclusions: A positive result (similar survival and prosthetic durability in group B, with lower complications) could change the current indications of AVS in our environment, allowing the age of indication of bioprostheses to be reduced below 60 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50-65 years who underwent isolated aortic valve replacement (AVR) for severe aortic stenosis from years 2000-2015 both inclusive

Exclusion Criteria:

* Not reported Residency change (unreachable)
* Need of concomitant surgery
* Reoperations
* Infective endocarditis

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 50-65 years who underwent isolated aortic valve replacement (AVR) for severe aortic stenosis from years 2000-2015 both inclusive, with bioprosthesis or mechanical prosthesis
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Number of participants alive | From date of surgery until the date of death from any cause, assessed up to 17 years
  Survival since surgery
Late postoperative endpoint of 4 MACE complications | From date of surgery until the date of first documented MACE (see description) or date of death from any cause, whichever came first, assessed up to 17 years
  All cause Mortality, major bleeding, cerebrovascular or transient ischemic accident, and need of any prosthesis reintervention (Major Adverse Cardiovascular Events, MACE)

SECONDARY OUTCOMES:
Total in-Hospital and Intensive Care Unit stay (in days) | From date of surgery to discharge of the unit and Hospital, up to 6 months
  Total in-Hospital and Intensive Care Unit stay (in days)
Cardiopulmonary bypass time in minutes needed in the surgery | day 1 after surgery
  Cardiopulmonary bypass time in minutes needed in the surgery
Cross-clamp ischemic heart time in minutes needed in the surgery | day 1 after surgery
  Cross-clamp ischemic heart time in minutes needed in the surgery
Transfusional requirements (number of red packed cells, fresh frozen plasma and platelets) | rom date of surgery until the date of first documented transfusional requirement assessed up to 17 years
  transfusional needs in long term follow up
Structural valve deterioration (SVD) in bioprosthesis | From date of surgery until the date of first documented SVD assessed up to 17 years
  increase in 20 mmHg in transaortic gradient since discharge echocardiography, any aortic regurgitation greater than moderate or need for bioprosthesis reoperation
Cardiovascular cause of rehospitalization | f first documented Cardiovascular cause of rehospitalization assessed up to 17 years
  any cardiovascular cause which need rehospitalization after surgery
Postsurgery Mean transprosthetic gradients in mmHg | From date of surgery until the date of Hospital Discharge, documented first Mean transprosthetic gradient in mmHg assessed by echocardiography after surgery.
  measured by the first echocardiography after surgery
Late Mean transprosthetic gradients in mmHg | From date of surgery until the date of last documented echocardiography assessed up to 17 years
  measured by the last echocardiography in follow up
Any prosthetic infective endocarditis | From date of surgery until the date of first documented prosthetic infective endocarditis, assessed up to 17 years
  definite diagnosis of early or late infective endocarditis

CONTACTS AND LOCATIONS:
Overall Officials: EMILIANO A RODRIGUEZ-CAULO, MD, PhD, Principal Investigator — FIMABIS, HOSPITAL VIRGEN DE LA VICTORIA DE MÁLAGA
Locations (7):
- Spain (7):
  - Hospital Regional Universitario de Malaga, Málaga, Málaga
  - Hospital Universitario Puerta Del Mar, Cadiz
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez-Caulo EA, Macias D, Adsuar A, Ferreiro A, Arias-Dachary J, Parody G, Fernandez F, Daroca T, Rodriguez-Mora F, Garrido JM, Munoz-Carvajal I, Barquero JM, Valderrama JF, Melero JM. Biological or mechanical prostheses for isolated aortic valve replacement in patients aged 50-65 years: the ANDALVALVE study. Eur J Cardiothorac Surg. 2019 Jun 1;55(6):1160-1167. doi: 10.1093/ejcts/ezy459. PMID 30608571